CLINICAL TRIAL: NCT05787236
Title: Moderate-to-severe Plaque Psoriasis Patients Response to Secukinumab Treatment in Real-world Setting: a Monocentric, Retrospective Study
Brief Title: A Study of Moderate-to-severe Plaque Psoriasis Patients Response to Secukinumab Treatment in Real-world Setting
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457AID01
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Moderate-to-severe Plaque Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Secukinumab: Clinical psoriasis patients who received secukinumab treatment in Indonesia from 1 August 2017 to 31 October 2020.

SUMMARY:
This study was a one-arm, retrospective cohort study that observed clinical psoriasis patients who received secukinumab treatment in Indonesia from the 01 August 2017 until the 31 October 2020. Patients' data were obtained from the medical records of a dermatology clinic in Jakarta, Indonesia. The primary endpoints were set at Week 16, and secondary endpoints at Weeks 16 and 52. At each endpoint, the study assessed effectiveness by measuring the proportion of psoriasis patients receiving secukinumab who achieved Psoriasis Area and Severity Index (PASI) 75 (at Week 8) and PASI 90 (at Weeks 16 and 52).

ELIGIBILITY:
Inclusion Criteria

* Male or female, aged at least 18 years old.
* Diagnosed as moderate-to-severe plaque type psoriasis with PASI score ≥ 5 prior to initiating secukinumab treatment.
* Treated with secukinumab for a minimum of 8 weeks after the initial secukinumab treatment without any interruption.
* Patients included in this study received the initial secukinumab treatment within the period of 1 August 2017 to 31 October 2019. With the secondary endpoint of 52 weeks, the latest recorded data included in the analysis was recorded on 31 October 2020.

Exclusion Criteria

* Patients with other types of psoriasis.
* Patients with incomplete information on PASI score at Weeks 0, 8, and 16 in their medical records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving Psoriasis Area and Severity Index (PASI) score <1, PASI score < 2, PASI score < 3, and PASI score < 5 at Week 16 | Week 16
  The PASI is used for assessing and grading the severity of psoriatic lesions and their response to therapy. PASI scores can range from a lower value of 0, corresponding to no signs of psoriasis, up to a theoretic maximum of 72.0.

SECONDARY OUTCOMES:
Percentage of patients achieving PASI 75 or higher response at Week 8 | Week 8
  PASI 75 response was defined as ≥ 75% improvement (reduction) in PASI score compared to baseline.
Percentage of patients achieving PASI 90 or higher response at Week 16 | Week 16
  PASI 90 response was defined as ≥ 90% improvement (reduction) in PASI score compared to baseline.
Percentage of patients achieving PASI 90 or higher response at Week 52 | Week 52
  PASI 90 response was defined as ≥ 90% improvement (reduction) in PASI score compared to baseline.
Number of injections needed to achieve at least PASI 90 | Weeks 16 and 52
  PASI 90 response was defined as ≥ 90% improvement (reduction) in PASI score compared to baseline.
Percentage of patients with psoriatic arthritis (PsA) who achieved at least PASI 90 at Week 16 with secukinumab | Week 16
  PASI 90 response was defined as ≥ 90% improvement (reduction) in PASI score compared to baseline.
Percentage of patients with relapse event after treatment discontinuation | Up to 52 weeks
Length of remission period for patients with relapse, calculated from the last treatment date until relapse or starting recurrent symptom(s) or sign(s) | Up to 52 weeks
Percentage of patients achieving Dermatology Life Quality Index (DLQI) 0/1 at Week 52 | Week 52
  DLQI is a ten-item general dermatology disability index designed to assess healthrelated quality of life in adult participants with skin diseases such psoriasis. It is a selfadministered questionnaire which includes domains of daily activity, leisure, personal relationships, symptoms and feelings, treatment and school/work activities. Each domain has 4 response categories ranging from 0 (not at all) 1 ( a little) to 3 (very much). "Not relevant" is a valid score also and is scored as 0.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Mangga Besar Clinic, Jakarta, Indonesia